CLINICAL TRIAL: NCT04567472
Title: HEADS: UP (Helping Ease Anxiety and Depression Following Stroke) Online Psychological Self-management Intervention: Feasibility Trial
Brief Title: HEADS: UP Online Psychological Self-management Intervention: Feasibility 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HLS/NCH/19/061
Record Dates: First submitted 2020-09-08; First posted 2020-09-28 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Stroke; CVA (Cerebrovascular Accident); Anxiety; Depression
Keywords: Stroke; CVA; Anxiety; Depression; Mindfulness; MBSR; Online; Self-management
MeSH Terms: conditions — Stroke; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online HEADS: UP (Experimental): HEADS: UP online is a group-based mindfulness course with an accompanying text-based manual. HEADS: UP comprises 9 x 2.5 hour mindfulness sessions, which incorporate a 30-minute break. A 6-hour silent retreat is offered in week 7. A follow-up session will be offered 6 - 8 weeks after the end of the course. Course materials include accessible information packs delivered weekly, electronically, and CD/audio resources to complement the sessions. The accompanying text-based manual will be delivered 'up front' (hard copy and electronic). A summary email and reminder of personal practice will be sent to participants after each session, including links to audio resources complementing class-based sessions. Signposting to other resources and media, including sites with downloadable voice files e.g. Mindfulness Scotland will be included.
  Interventions: Behavioral: Helping Ease Anxiety and Depression following Stroke

INTERVENTIONS:
Behavioral: Helping Ease Anxiety and Depression following Stroke — HEADS: UP online is a group-based mindfulness course with an accompanying text-based manual. HEADS: UP comprises 9 x 2.5 hour mindfulness sessions, which incorporate a 30-minute break. A 6-hour silent retreat is offered in week 7. A follow-up session will be offered 6 - 8 weeks after the end of the course. Course materials include accessible information packs delivered weekly, electronically, and CD/audio resources to complement the sessions. The accompanying text-based manual will be delivered 'up front' (hard copy and electronic). A summary email and reminder of personal practice will be sent to participants after each session, including links to audio resources complementing class-based sessions. Signposting to other resources and media, including sites with downloadable voice files e.g. Mindfulness Scotland will be included.
  Other Names: HEADS: UP

SUMMARY:
To test feasibility of online version of HEADS: UP

DETAILED DESCRIPTION:
Study aim(s): to conduct feasibility testing of online HEADS: UP, a tailored adaptation of an existing psychological intervention (MBSR) to help people affected by stroke self-manage symptoms of anxiety and depression.

Objectives: 1) Assess feasibility and acceptability of delivering the HEADS: UP intervention online and identify any additional adaptations to the HEADS: UP manual and supporting materials. 2) Assess feasibility and acceptability of online research processes, including recruitment, screening, and obtaining informed consent, and data collection processes.

Research question: What elements of intervention design, delivery, and study processes require to be optimised ahead of a 3-arm RCT?

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Have had ≥1 stroke at least 3 months previously
* Interested in learning skills to help cope with self-reported anxiety and/or depression
* Able to speak and understand conversational English
* Score ≥ 4 on either sub-scale Hospital Anxiety and Depression Scale (HADS)
* Desirable: Able to identify a family member/peer who would: like to take part, can speak and understand conversational English; not participating in another trial.

Potential participants who do not identify someone else to take part with them will not be excluded.

Exclusion Criteria:

* Prior MBSR attendance in the last three years (as this may confound results)
* Current participant in another trial
* Cannot follow a 2-stage command

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory II (BDI-II): change is being assessed | Weeks 0, 9
  The Beck Depression Inventory 11 (BDI-II) is a 21 items self-report scale to assess the intensity of depression. Each item is a list of four statements arranged in increasing severity about a symptom of depression. Score range between 0-63 with higher score indicating greater severity. Normally completed in 5-10 minutes.
Beck Anxiety Inventory (BAI): change is being assessed | 0, 9 weeks
  The Beck Anxiety Inventory (BAI) is a self-report 21-item scale for measuring anxiety. The questions ask about symptoms of anxiety the subject has had during the past week. Each question is scored between 0 (mild) and 3 (severe) and a total score will vary between 0-63. Higher scores indicate more severe anxiety symptoms.
. Depression Anxiety Stress Scale (DASS): change is being assessed | Weeks 0, 9
  The DASS is a set of three self-report scales designed to measure depression, anxiety and stress. Each of the three DASS scales contains 14 items, divided into subscales of 2-5 items with similar content. The Depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia. The Anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The Stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient. Subjects are asked to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items.
EQ-5D 5L: change is being assessed | Weeks 0, 9
  The 5-level EQ-5D version (EQ-5D-5L) comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Stroke Impact Scale (SIS): change is being assessed | Weeks 0, 9
  The Stroke Impact Scale (SIS) is a self-report, health status measure for people affected by stroke. It was designed to assess strength, hand function, activities of daily living, mobility, communication, emotion, memory and thinking, and participation. The SIS can be used both in clinical and research settings. It contains 59 items and assesses 8 domains. Each item is rated using a 5-point Likert scale. A final single-item question assesses the individual's perception of recovery from stroke, measured using a visual analogue scale, where 0 = no recovery & 100 = full recovery. The scale is normally completed in 15-20 minutes.
Focus group | Week 9
  Focus Groups (FGs) will be used to collect qualitative data.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Lawrence, Dr., Study Director — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, Glasgow (City Of), United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HELPING EASE ANXIETY AND DEPRESSION AFTER STROKE (HEADS: UP) — https://www.cso.scot.nhs.uk/wp-content/uploads/HIPS1663RPB.pdf